CLINICAL TRIAL: NCT03296878
Title: Food-for-Families: Relationship Between Income, Obesity, and Food Purchasing Using an Experimental Grocery Store Study
Brief Title: Food-for-Families: Experimental Grocery Store Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: GFHNRC151
Record Dates: First submitted 2017-09-25; First posted 2017-09-28 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Overweight; Obesity
Keywords: low income
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: This study will utilize a three factor design, with one between-subject factor and two within-subject factors. The between-subject factor is participation in a federal food assistance program. The within-subject factors are price change condition and price change scenario.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Own-Price Elasticity (Other): The price of eggs will vary (own-price elasticity) while the price of other foods in the "mock" grocery store will remain constant.
  Interventions: Other: Own-Price Elasticity
- Cross-Price Elasticity (Other): The eggs will remain constant while the price of other foods in the "mock" grocery store will vary (cross-price elasticity).
  Interventions: Other: Cross-Price Elasticity

INTERVENTIONS:
Other: Own-Price Elasticity — The price of eggs will be 75%, 100%, or 125% of the reference price, but the price of other foods will remain the same.
  Arms: Own-Price Elasticity
Other: Cross-Price Elasticity — The price of eggs will remain the same, but the price of other foods will be 75%, 100%, or 125% of the reference price.
  Arms: Cross-Price Elasticity

SUMMARY:
This is a study about how the price of foods affects buying choices at the grocery store. The price of foods can have a big impact on what people choose to buy and prices change over time. This study is being done to see how changes in food prices affect what mothers choose for their families.

DETAILED DESCRIPTION:
It is well known that the price of a given food affects the amount of that item individuals will purchase. Yet little is known about how specific groups, such as obese/overweight individuals and those with lower incomes, change their food purchasing decisions depending on food price changes. Evidence shows that these groups have lower quality diets and worse health outcomes than their normal weight and higher income counterparts. Therefore, it is important to gain a better understanding of how food price changes affect purchasing decisions among these population groups in order to develop targeted nutrition interventions to improve their diet quality. To investigate this, the researchers will create a laboratory-based grocery store, in which pictures of foods will be used in lieu of actual foods. Food prices will be indicated on each picture. The participants will be given play money and a budget, and asked to "purchase" foods in the mock grocery store. The price of foods will be changed throughout the study to investigate how participants change their purchasing decisions based on these price changes.

ELIGIBILITY:
Inclusion Criteria:

* Have at least one child up to 18 years of age residing in the household
* Primary grocery shopper for the household
* No health conditions or food practices that substantially limit food choice
* Not currently pregnant
* Consent to the study design

Exclusion Criteria:

* Male
* < 18 years of age
* Not a mother, or children not living with subject in their household
* No children below the age of 18 years of age
* Not the primary grocery shopper for their household
* Health conditions or food practices that substantially limit food choice
* Currently pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Price elasticity of eggs | Baseline
  Percent change in the amount of eggs purchased (gram weight) for every percent change in the price of a given food.

SECONDARY OUTCOMES:
Nutrient density of purchased foods | Baseline
  Ratio of low nutrient-dense food purchases to high nutrient-dense food purchases

CONTACTS AND LOCATIONS:
Overall Officials: James Roemmich, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No